CLINICAL TRIAL: NCT03635606
Title: Validation of AKI-Sapere Model to Predict Patients at Risk for AKI After Cardiac Surgery: GUARD-AKI (GUiding Against Reserve Decline)
Brief Title: GUARD-AKI: Validation of AKI-Sapere in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Sapere Bio (Industry)
Collaborators: WakeMed Health and Hospitals (Other); Johns Hopkins University (Other); Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Other Study IDs: HSDX-1801
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac surgery associated acute kidney injury (CSA-AKI) has been recognized as the second most common cause of hospital acquired AKI. The development of CSA-AKI is independently associated with an increased risk of in-hospital death. There are currently no biomarkers that could identify patients at higher risk for AKI and current risk predictor scores that are based on clinical and demographic information are inadequate. Therefore, a diagnostic test for predicting AKI risk in this clinical context would assist clinicians to optimize surgical strategy and postoperative care to prevent CSA-AKI occurrence and improve patient outcomes.

The primary purpose of this study is to validate a panel of biomarkers identified in the discovery study (referred to as AKI-Sapere prognostic) to identify patients at risk for all stages of CSA-AKI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>40 years) undergoing non-emergency (urgent or scheduled) cardiac surgery using cardiopulmonary bypass (CABG or combined CABG/valve).
* Patients must be able to understand English and be willing to sign informed consent.

Exclusion Criteria:

* Emergency surgery
* Off-pump coronary bypass grafting
* Aortic aneurysm repair
* Congenital heart disease repair
* Heart transplant or left ventricular assist device patient
* Severe heart failure (left ventricular ejection fraction <25%)
* Hemodynamic instability or requiring preoperative vasopressors or IABP
* Pre-existing kidney disease (eGFR <30 mL/min/1.73 m2) or renal transplantation.
* Presence of major active infection (chronic or acute, eg, sepsis, HIV, pneumonia)
* Chronic liver disease/cirrhosis
* Participation in an additional trial at the time of surgery or anytime within 30d of surgery where intervention could potentially alter renal health (unless in the control arm)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects entered into this study will be patients at the participating institutions.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Development of stage 1 or higher postoperative AKI as defined by the KDIGO classification (stage 1 = sCr value of ≥0.3 mg/dL in the first 48h or a relative increase of ≥50% in peak sCr from baseline within 7 days post-surgery) | within 7 days post-surgery

SECONDARY OUTCOMES:
Development of moderate to severe AKI (sCr increase of ≥100% within 7 days post surgery or a sCr increase of ≥100% from baseline within 7 days and urine output <0.5 mL/kg/h for >12h) | within 7 days post-surgery
Development of 30-day persistent kidney impairment (eGFR change of ≥25% from baseline at the 30-day follow-up visit) | 30 days post-surgery
Development of new onset atrial fibrilation | within 7 days post-surgery
Development of 30-day major adverse kidney events (MAKE30): a composite of persistently impaired renal function (sCr increase of ≥0.5 mg/dL from baseline [pre-surgery]), new dialysis, and death | 30 days post-surgery
Development of 30-day major adverse cardiac events (MACE30): a composite of myocardial infarction (MI), stroke, heart failure, and death | 30 days post-surgery
Development of the combination of MAKE30 and MACE30 (major adverse reno-cardiovascular events [MARCE30]) | 30 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Mitin, PhD, Principal Investigator — Sapere Bio
Locations (3):
- United States (3):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Johns Hopkins University, Baltimore, Maryland
  - WakeMed Health and Hospitals, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No